CLINICAL TRIAL: NCT03323593
Title: Crossover Pharmacokinetic Study of Two Mode of Administration of Intranasal Dexmedetomidine in Healthy Adult Volunteers
Brief Title: Pharmacokinetics of Different Mode Administration of Intranasal Dexmedetomidine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, YUEN, Vivian Man-ying, Dr, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PK InDexm
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Bioavailability; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- iv (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- drip (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- atomizer (Active Comparator)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — blood is sampled for quantification of plasma concentration after intravenous, intranasal by atomisation and intranasal by drops.

SUMMARY:
Intranasal dexmedetomidine has been studied and used in children for premedication before anaesthesia or fro sedation. It can be administered by simple dripping or by Mucosal Atomization Device (MAD®).

Since MAD® delivers intranasal medication in a fine mist, it is possible that absorption and bioavailability would be better compares to simple dripping method. To date no pharmacokinetic information of intranasal dexmedetomidine delivered by either method is available. This investigation is designed to compare the bioavailablity of intranasal dexmedetomidine deliver via simple dipping with tuberculine syringe and MAD® in healthy adults.

DETAILED DESCRIPTION:
This is a three-period crossover double-blinded study. 8 subjects will be recruited and they will attend 3 study sessions after informed written and verbal consent. They would have dexmedetomidine administered via different rout each time, intravenous, intranasal via dripping or intranasal via atomizer. Blood samples are collect to determine bioavailability of each mode of drug delivery.

ELIGIBILITY:
Inclusion Criteria:

healthy volunteer ASA 1 age over 18 no other concomitant drug therapy no alcohol or smoking habit -

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Bioavailability of dexmedetomidine | 8 hours

SECONDARY OUTCOMES:
sedation score | 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong